CLINICAL TRIAL: NCT05833035
Title: A Phase I, Open-label, Single Dose, Mass Balance Trial to Investigate Metabolism and Pharmacokinetics of BI 1291583 (C-14) Administered as Oral Solution in Healthy Male Subjects
Brief Title: A Study in Healthy Men to Test How BI 1291583 is Processed in the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1397-0016
Record Dates: First submitted 2023-04-17; First posted 2023-04-27 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2024-06

CONDITIONS: Healthy
MeSH Terms: interventions — Carbon-14

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BI 1291583 (C-14) (Experimental)
  Interventions: Drug: BI 1291583 mixed with [C-14] BI 1291583

INTERVENTIONS:
Drug: BI 1291583 mixed with [C-14] BI 1291583 — BI 1291583 mixed with radioactive carbon labelled [C-14] BI 1291583

SUMMARY:
The main objective of this trial is to

* Assess the mass balance and total recovery of [14C]-radioactivity in urine and faeces following a dose of BI 1291583 (C-14)
* Provide plasma and urine samples for pharmacokinetic investigations
* Provide plasma, urine, and faeces samples for metabolic profiling and structural identification of metabolites

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kilogram per square meter (kg/m2, inclusive)
* Signed and dated written informed consent in accordance with International Council for Harmonization - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimeter of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ICON, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was performed as an open-label, single-arm, single-dose trial in healthy male subjects to investigate the basic PK of BI 1291583, its metabolites (BI 1373234, CD 18507, CD 17849, CD 16785, and BI 1321869 (CD 16426)) and [14C]-radioactivity, including mass balance, excretion pathways and metabolism following a single oral dose of 5 mg BI 1291583 (C-14).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that the subjects strictly met all inclusion and none of the exclusion criteria. Subjects were not to be entered in the trial if any of the entry criteria were violated.
Groups:
- BI 1291583 (C-14): Participants received a single dose of 20 milliliter (mL) of BI 1291583 (C-14) radioactive solution for oral administration concentrated at 0.25 milligram/mL. The radioactive solution contained a radioactive dose of approximately 0.36 Megabecquerel (MBq). The oral solution contained a mixture of pure radioactive carbon [14C]-labelled "hot" drug substance, and BI 1291583, i.e. unlabelled "cold" drug substance. The BI 1291583 (C-14) oral solution was administered with 240 mL of water after an overnight fast of at least 10 hours (h).
Period: Overall Study
Arm/Group | BI 1291583 (C-14)
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): included all subjects who were treated with at least one dose of trial drug.
Arm/Group | BI 1291583 (C-14)
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mass Balance and Total Recovery of [14C]-Radioactivity in Urine: Fraction of [14C]-Radioactivity Excreted in Urine Expressed as Percentage of the Administered Dose Over the Time Interval From 0 to the Last Quantifiable Time Point (Feurine, 0-tz)
Description: Fraction of [14C]-radioactivity excreted in urine expressed as percentage of the administered dose over the time interval from 0 to the last quantifiable time point (feurine, 0-tz) is reported.
  Timeframe: After 336h, 24h interval urine sample collection was planned every 7 days starting on Day 21 until Day 43.
Time Frame: Urine sampling intervals: Within 14 hours (h) prior and 0-4 , 4-8, 8-12, 12-24, 24-48, 48-72, 72-96, 96-120, 120-144, 144-168, 168-192, 192-216, 216-240, 240-264, 264-288, 288-312, 312-336h after intake of BI 1291583 (C14). Continues in description.
Population: Pharmacokinetic set (PKS): This set included all subjects in the treated (TS) who provided at least one pharmacokinetic (PK) endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject was included in the PKS, even if he/she contributed only one PK parameter value for one period to the statistical assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of administered dose
Arm/Group | BI 1291583 (C-14)
Number analyzed (Participants) | 8
percentage of administered dose | 26.0 (12.9)

2. Primary Outcome: Mass Balance and Total Recovery of [14C]-Radioactivity in Faeces: Fraction of [14C]-Radioactivity Excreted in Faeces Expressed as Percentage of the Administered Dose Over the Time Interval From 0 to the Last Quantifiable Time Point (Fefaeces, 0-tz)
Description: Fraction of [14C]-radioactivity excreted in faeces expressed as percentage of the administered dose over the time interval from 0 to the last quantifiable time point (fefaeces, 0-tz) is reported.
  Timeframe: After 336h, 24h interval stools sample collection was planned every 7 days starting on Day 21 until Day 43.
Time Frame: All stools were collected prior and up to 336 hours (h) (sampling intervals 0-24, 24-48, 48-72, 72-96, 96-120, 120-144, 144-168, 168-192, 192-216, 216 -240, 240-264, 264-288, 288-312, 312-336 h) after intake of BI 1291583 (C14). Continues in description.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of administered dose
Arm/Group | BI 1291583 (C-14)
Number analyzed (Participants) | 8
percentage of administered dose | 61.4 (13.2)

3. Secondary Outcome: Area Under the Concentration-time Curve of [14C]-Radioactivity ([14C]-BI 1291583-Equivalents (EQ)) in Plasma Over the Time Interval From 0 to the Last Quantifiable Time Point (AUC0-tz, [14C]-BI 1291583-EQ)
Description: Area under the concentration-time curve of [14C]-radioactivity ([14C]-BI 1291583-EQ) in plasma over the time interval from 0 to the last quantifiable time point (AUC0-tz, [14C]-BI 1291583-EQ) is reported.
Time Frame: Within 4 hours prior and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 24, 48, 72, 120, 168, 216, 264, 336, 485, 653, 821, 989 hours after administration of BI 1291583 (C14).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour * nanomole/Liter (h*nmol/L)
Arm/Group | BI 1291583 (C-14)
Number analyzed (Participants) | 8
hour * nanomole/Liter (h*nmol/L) | 1730 (16.1)

4. Secondary Outcome: Area Under the Concentration-time Curve of BI 1291583 in Plasma Over the Time Interval From 0 to the Last Quantifiable Time Point (AUC0-tz, BI 1291583)
Description: Area under the concentration-time curve of BI 1291583 in plasma over the time interval from 0 to the last quantifiable time point (AUC0-tz, BI 1291583) is reported.
Time Frame: Within 4 hours (h) prior and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 24, 48, 72, 120, 168, 216, 264, 336, 485, 653, 821, 989 h after administration of BI 1291583 (C14).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour * nanomole/Liter (h*nmol/L)
Arm/Group | BI 1291583 (C-14)
Number analyzed (Participants) | 8
hour * nanomole/Liter (h*nmol/L) | 139 (19.7)

5. Secondary Outcome: Maximum Measured Concentration of [14C]-Radioactivity ([14C]-BI 1291583-Equivalents (EQ)) in Plasma (Cmax, [14C]-BI 1291583-EQ)
Description: Maximum measured concentration of [14C]-radioactivity ([14C]-BI 1291583-EQ) in plasma (Cmax, [14C]-BI 1291583-EQ) is reported.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter (nmol/L)
Arm/Group | BI 1291583 (C-14)
Number analyzed (Participants) | 8
nanomole/Liter (nmol/L) | 6.58 (14.4)

6. Secondary Outcome: Maximum Measured Concentration of BI 1291583 in Plasma (Cmax, BI 1291583)
Description: Maximum measured concentration of BI 1291583 in plasma (Cmax, BI 1291583) is reported.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter (nmol/L)
Arm/Group | BI 1291583 (C-14)
Number analyzed (Participants) | 8
nanomole/Liter (nmol/L) | 1.90 (23.8)

7. Secondary Outcome: Area Under the Concentration-time Curve of BI 1291583 Metabolites in Plasma Over the Time Interval From 0 to the Last Quantifiable Time Point (AUC0-tz, BI 1291583 Metabolites)
Description: Area under the concentration-time curve of BI 1291583 metabolites in plasma over the time interval from 0 to the last quantifiable time point (AUC0-tz, BI 1291583 metabolites). AUC0-tz of the following BI 1291583 metabolites is reported:
  BI 1373234; CD 18507; CD 17849; CD 16785; BI 1321869.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour *nanomole/Liter (h*nmol/L)
Arm/Group | BI 1291583 (C-14)
Number analyzed (Participants) | 8
hour *nanomole/Liter (h*nmol/L)
  CD 17849 | 157 (47.8)
  CD 18507 | 159 (37.3)
  CD 16785 | 167 (47.6)
  BI 1373234 | 48.3 (33.2)
  BI 1321869 | 5280 (79.4)

8. Secondary Outcome: Maximum Measured Concentration of BI 1291583 Metabolites in Plasma (Cmax, BI 1291583 Metabolites)
Description: Maximum measured concentration of BI 1291583 metabolites in plasma (Cmax, BI 1291583 metabolites). Cmax of the following metabolites is reported:
  BI 1373234; CD 18507; CD 17849; CD 16785; BI 1321869.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter (nmol/L)
Arm/Group | BI 1291583 (C-14)
Number analyzed (Participants) | 8
nanomole/Liter (nmol/L)
  CD 17849 | 1.48 (44.9)
  CD 18507 | 0.944 (28.3)
  CD 16785 | 0.330 (43.6)
  BI 1373234 | 0.391 (26.3)
  BI 1321869 | 12.2 (26.2)

ADVERSE EVENTS:
Time Frame: From first administration of BI 1291583 (C14) until the end of the residual effect period, up to 28 days.
Description: Treated set (TS): included all subjects who were treated with at least one dose of trial drug.
Arm/Group | BI 1291583 (C-14)
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 5/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1291583 (C-14) (N=8)
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/35/NCT05833035/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT05833035/SAP_001.pdf